CLINICAL TRIAL: NCT04386408
Title: Preliminary Study on the Effect of Consuming a Combination of Plant Extracts (BSL_EP027) on the Incidence of Respiratory Infection Symptoms in Healthy Elderly Living in a Nursing Home.
Brief Title: Evaluation of the Effect of a Combination of Plant Extracts (BSL_EP027) on the Incidence of Respiratory Infections
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biosearch S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C027
Record Dates: First submitted 2019-11-14; First posted 2020-05-13 (Actual); Last update posted 2020-05-13 (Actual); Status verified 2019-07

CONDITIONS: Immune Response; Respiratory Diseases
Keywords: Immunostimulation; Respiratory diseases; Plant extracts
MeSH Terms: conditions — Respiratory Tract Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Combination of plant extracts (BSL_EP027) (Experimental): Volunteers will dissolve in water a sachet per day with the Combination of plant extracts (BSL_EP027), and maltodextrin.
  Interventions: Combination Product: Combination of plant extracts (BSL_EP027)
- Placebo (Placebo Comparator): Volunteers will dissolve in water a sachet per day with maltodextrin.
  Interventions: Combination Product: Placebo

INTERVENTIONS:
Combination Product: Combination of plant extracts (BSL_EP027) — Each participant will consume a sachet disolve in water once at day without any restriction in the diet nor in their habits of life.
  Arms: Combination of plant extracts (BSL_EP027)
Combination Product: Placebo — Each participant will consume a sachet disolve in water once at day without any restriction in the diet nor in their habits of life.
  Arms: Placebo

SUMMARY:
The objective of the present study is to evaluate the effectiveness of daily consumption of a Combination of Plant Extracts (BSL_EP027) on the incidence of respiratory infection symptoms and their duration in older healthy volunteers living in a nursing home.

DETAILED DESCRIPTION:
A prevalence of deficient immune state is estimated at 44% of the world's population, a figure that rises in the senior population group.

Traditionally, protection against infection and improvement of the immune response has been addressed through the use of plant extracts. An effective immune response involves the action of both innate and specific responses and the perfect coordination between both. Natural strategies that can activate both types of immune response can lead to more effective treatments.

Our hypothesis is that the different effects of the combination of several plant extracts can lead to a synergy that generates a more effective product in the prevention of respiratory infections, especially in susceptible populations such as the elderly.

ELIGIBILITY:
Inclusion Criteria:

* Living in a nursing home with medical service.
* Freely accept to participate in the study and sign the informed consent document.

Exclusion Criteria:

* Having a disease that affects the development and results of the study.
* Suffer alterations of the state of health incompatible with the continuity in the study.
* Suffer any adverse event not tolerated by the subject.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-11-30 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
Respiratory infection symptoms | 16 weeks
  Incidence of respiratory infection symptoms (fiber, cough, rinitis, headache, sore throat, bone and/or muscle pain, fatigue/exhaustion, nausea and/or vomiting, lack of appetite and /or trouble for sleeping)

SECONDARY OUTCOMES:
Duration of the respiratory infection symptoms | 16 weeks
  Duration of the respiratory infection symptoms (days)

OTHER OUTCOMES:
Type of Medication for the respiratory infection symptoms | 16 weeks
  Type of medication for the respiratory infection symptoms
Dose of the Medication for the respiratory infection symptoms | 16 weeks
  Dose of the medical treatment for the respiratory infection symptoms
Duration of the medical treatment for the respiratory infection symptoms | 16 weeks
  Duration of the medical treatment for the respiratory infection symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Gracián, MD, Principal Investigator — Doctor of the Claret Nursing Home (Granada, Spain)
Locations (1):
- Claret Nursing home, Granada, Spain

IPD SHARING:
Plan to Share IPD: No